CLINICAL TRIAL: NCT01542593
Title: Evaluation of Ureteral Length Measurement by Computed Tomography (CT) to Actual Ureteral Length Measured by Ureteral Catheterization
Brief Title: Evaluating Ureteral Length Using Computed Tomography (CT)
Acronym: URO-Y-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Yuval Freifeld, Resident , Urology Department, principal investigator, Medical doctor, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-11-0051-CTIL
Record Dates: First submitted 2012-02-16; First posted 2012-03-02 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Ureteral Calculi; Hydronephrosis; Ureteral Obstruction
MeSH Terms: conditions — Ureteral Calculi; Hydronephrosis; Ureteral Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ureteral catheterization (Experimental): During a planned procedure involving ureteroscopy or ureteral stenting, ureteral catheterization will be performed for the purpose of measuring exact ureteral length.
  Measurement results will be compared to measurements performed on CT scan (obtained before surgery).
  Interventions: Device: Ureteral catheterization - Cook Urological Inc. open end ureteral catheter 5FR

INTERVENTIONS:
Device: Ureteral catheterization - Cook Urological Inc. open end ureteral catheter 5FR — During a planned procedure involving ureteroscopy or ureteral stenting, after retrograde pyelography and insertion of a safety wire, ureteral catheterization will be performed using Cook Urological Inc. open end ureteral catheter 5FR for the purpose of measuring exact ureteral length.
  Measurement results will be compared to measurements performed on CT scan (obtained before surgery).
  Other Names: Cook Urological Inc. open end ureteral catheter 5FR; Karl Storz cystoscope 19-22F

SUMMARY:
Proper selection of ureteral stent length might help in reducing comorbidities associated with ureteral stenting, currently there is no standardized way of measuring ureteral length.

Measurement of ureteral length according to Computed Tomography (CT) scan might provide useful information when selecting the length of a ureteral stent. Our aim in this study is to compare ureteral measurements using CT scan and measurement of actual ureteral length measured during ureteral stenting.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing planned procedure involving ureteroscopy or ureteral stenting
* Abdominal CT scan performed within 6 months prior to intervention

Exclusion Criteria:

* Known iodine sensitivity
* Patients with fever or hemodynamic instability planned for urgent operation
* Severe immune compromized patients
* Severe thrombocytopenia < 50,000

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Agreement between measurement of ureteral length (Centimeters) measured by CT and by ureteral catheterization | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Freifeld, Dr., Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel